CLINICAL TRIAL: NCT07371975
Title: A Study to Evaluate the Effects of a Butyrate-Polyphenol Formulation on Gut Health and Associated Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Supplement Formulators, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL116
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Gut Health
Keywords: Gastrointestinal discomfort; Abdominal pain; Gas; Bloating; Diarrhea; Constipation
MeSH Terms: conditions — Abdominal Pain; Mucopolysaccharidosis IV; Diarrhea; Constipation | interventions — Butyrates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butyrate + Polyphenol Formulation (Active Comparator): Butyrate + Polyphenol Formulation
  Interventions: Dietary Supplement: Butyrate + Polyphenol Formulation
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Butyrate + Polyphenol Formulation — Butyrate + Polyphenol Formulation
  Arms: Butyrate + Polyphenol Formulation
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy of a butyrate/polyphenol formulation on modulation of the gut microbiome and gastrointestinal symptoms using questionnaires in individuals with self-reported gastrointestinal discomfort.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled study to evaluate the effects of a butyrate/polyphenol formulation on gut health and associated symptoms in healthy individuals.

Participants will be asked to complete a laboratory assessment and questionnaires. A total of up to 124 subjects (62 subjects per arm) will be enrolled for the 14-day period. Laboratory testing will include an assessment of the Gut Microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 25-70 years
2. Body mass index 18.5-34.9 kg/m2
3. A GSRS-IBS score ≥ 21 (identification as having moderate or severe gastrointestinal symptoms). If the GSRS-IBS score is < 20 (identification of minimal or mild), may be included at the discretion of the PI/Sub-I
4. Experiencing at least three of the following conditions on a weekly basis (gastrointestinal discomfort, abdominal pain, gas, bloating, diarrhea, or constipation)
5. Healthy based on medical history and without chronic disease (unless permitted in the judgment of the PI/Sub-I)
6. Weight stable for the past six months (±6 lbs.)
7. Willing and able to give written informed consent
8. Ability to communicate and read in English
9. Ability to comply with study requirements

Exclusion Criteria:

1. Currently participating in another clinical research study
2. Pregnant, planning pregnancy, or breastfeeding
3. Unable to swallow capsules, tablets, or softgels
4. Male participants and females of childbearing potential who are unwilling to use an acceptable method of contraception from screening through 30 days after study completion.
5. Typically goes longer than 3 days without a bowel movement
6. Current diagnosis of cardiovascular disease, history of an abnormal electrocardiogram (ECG), diabetes (Type 1 or Type 2), or cancer (except for non-melanoma skin cancer) within the past 5 years
7. Having had a medical or surgical event in the past 5 years involving hospitalization, outpatient, or emergency care that requires ongoing monitoring.
8. Planning to undergo a major medical procedure or surgical event within the next 30 days
9. Currently being treated for any infectious disease
10. Currently consuming more than 6 standard alcoholic drinks per week for women and 10 drinks per week for men (a standard alcoholic drink is defined as one bottle/can of beer, one glass of wine, or one ounce of hard liquor)
11. Smoking or use of nicotine products daily within 30 days prior to screening
12. Using substances of abuse or recreational drugs/substances, including tetrahydrocannabinol (THC), within the past 14 days
13. History of intolerance or allergic reaction to product ingredients, including butyrate, tributyrin, polyphenols (Green tea extract, Grape Seed extract, Cinnamon extract, maltodextrin, silicon dioxide, magnesium stearate, or chlorophyllin)
14. Having donated blood or received a blood/plasma transfusion within 30 days before baseline
15. History of a major change in dietary habits within the past 1 month
16. Currently taking any supplements containing butyrate, tributyrin, or polyphenols and not willing to stop for the duration of study participation
17. Currently taking any laxatives on a daily basis
18. Initiated (Glucagon-Like Peptide-1) GLP-1 medication within 3 months prior to screening.
19. On a stable dose of a proton pump inhibitor (e.g., omeprazole, pantoprazole) within 3 months prior to screening.
20. History of oral or IV antibiotic use within the past 3 months prior to Baseline
21. Not willing to refrain from taking any over-the-counter medications or supplements for gastrointestinal concerns or discomfort (except if on a stable dose for > 3 months before Screening and unlikely to change) unless in the judgment of the PI/Sub-I
22. Current or previous history of medically diagnosed and treated gastrointestinal disease, including gallbladder problems, gallstones, biliary obstruction, inflammatory bowel disease (IBD), Crohn's disease, Ulcerative Colitis, Celiac disease, or gastrointestinal cancer
23. Currently diagnosed with and/or being treated for Irritable Bowel Syndrome (IBS)
24. Currently experiencing or previously having a gastrointestinal infection (viral or bacterial) or food poisoning within the past month
25. Currently experiencing or previously having a parasitic infection within the past 3 months
26. Currently experiencing or having a history of severe endometriosis
27. History of gastrointestinal surgery, which might influence gastrointestinal function
28. History or presence of a clinically significant diagnosis or circumstance that, in the judgment of the Study Investigator/Sub-I, would interfere with the interpretation of the study results and preclude participation in the study -

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-04-26 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
The Gastrointestinal Symptom Rating Scale (GSRS)-Irritable Bowel Syndrome (IBS) version | 14 days
  Change in the Gastrointestinal Symptom Rating Scale-IBS from baseline. The responses to the questions range from no discomfort at all to very severe discomfort which would indicate a worse outcome
Gut Microbiome Stool Test | 14 days
  Change in the Gut Microbiome (strain level, functional metrics, taxonomy abundance and composition) from baseline

SECONDARY OUTCOMES:
Digestion-Associated Quality of Life Questionnaire (DQLQ) | 14 days
  Change in the Digestion-Associated Quality of Life Questionnaire (DQLQ) from baseline. The lower score indicates an improved outcome.
Visual Analogue Scale (VAS) of abdominal pain | 14 days
  Change in the Visual Analogue Scale (VAS) of abdominal pain from baseline. The lower the value indicates an improved outcome.
Bristol Stool Form Scale (BSFS) | 14 days
  Change in the stool form from baseline. There are 7 various stool types to choose ranging from Type 1 to Type 7. Types 3 or 4 are the preferred types.
Gastrointestinal -Global Assessment of Improvement Scale (Gastrointestinal-GAI) | 14 days
  Change in the Gastrointestinal-Global Assessment of Improvement Scale (Gastrointestinal-GAI) from baseline. The responses range from substantially worse to substantially improved would indicate an improved outcome.
World Health Organization Quality of Life (WHOQOL-BREF) | 14 days
  Change in the World Health Organization Quality of Life (WHOQOL-BREF) from baseline. The higher score indicates a better perceived quality of life for each domain.(physical health, psychological health, social relationship, environment)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Swick, PhD, Principal Investigator — Life Extension
Locations (1):
- Life Extension Clinical Research, Inc., Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Administration, D. o. H. a. H. S. U. S. F. a. D. (2005). Guidance for industry : estimating the maximum safe starting dose in initial clinical trials for therapeutics in adult healthy volunteers : pharmacology and toxicology. Center for Drug Evaluation and Research.
- [Background] Cleophas MCP, Ratter JM, Bekkering S, Quintin J, Schraa K, Stroes ES, Netea MG, Joosten LAB. Effects of oral butyrate supplementation on inflammatory potential of circulating peripheral blood mononuclear cells in healthy and obese males. Sci Rep. 2019 Jan 28;9(1):775. doi: 10.1038/s41598-018-37246-7. PMID 30692581
- [Background] Conley BA, Egorin MJ, Tait N, Rosen DM, Sausville EA, Dover G, Fram RJ, Van Echo DA. Phase I study of the orally administered butyrate prodrug, tributyrin, in patients with solid tumors. Clin Cancer Res. 1998 Mar;4(3):629-34. PMID 9533530
- [Background] Cory H, Passarelli S, Szeto J, Tamez M, Mattei J. The Role of Polyphenols in Human Health and Food Systems: A Mini-Review. Front Nutr. 2018 Sep 21;5:87. doi: 10.3389/fnut.2018.00087. eCollection 2018. PMID 30298133
- [Background] Costa C, Tsatsakis A, Mamoulakis C, Teodoro M, Briguglio G, Caruso E, Tsoukalas D, Margina D, Dardiotis E, Kouretas D, Fenga C. Current evidence on the effect of dietary polyphenols intake on chronic diseases. Food Chem Toxicol. 2017 Dec;110:286-299. doi: 10.1016/j.fct.2017.10.023. Epub 2017 Oct 14. PMID 29042289
- [Background] Cristofori F, Calabrese FM, Iacobellis I, Santamaria M, Celano G, Ferrocino I, Di Sabato E, Pergola R, Dargenio VN, Paulucci L, De Angelis M, Francavilla R. Calcium butyrate efficacy in pediatric irritable bowel syndrome: Randomized placebo-controlled multiomics-based clinical trial. J Pediatr Gastroenterol Nutr. 2025 Sep;81(3):551-561. doi: 10.1002/jpn3.70154. Epub 2025 Jul 9. PMID 40635319
- [Background] Grosicki, G. (2021). Effects of 3-week Tributyrin Supplementation on the Gut Microbiome: A Pilot Study. Journal of the Academy of Nutrition and Dietetics, 121(9), A23.
- [Background] Hodges, J. Z., M.; Cao, S.; Pokala, A.; Rezaei, S.; Sasaki, G.; Vodovotz, Y.; Bruno, R. (2022). Catechin-Rich Green Tea Extract Reduced Intestinal Inflammation and Fasting Glucose in Metabolic Syndrome and Healthy Adults: A Randomized, Controlled, Crossover Trial. Current Developments in Nutrition, 6, 981. https://doi.org/10.1093/cdn/nzac068.010
- [Background] Hodgkinson K, El Abbar F, Dobranowski P, Manoogian J, Butcher J, Figeys D, Mack D, Stintzi A. Butyrate's role in human health and the current progress towards its clinical application to treat gastrointestinal disease. Clin Nutr. 2023 Feb;42(2):61-75. doi: 10.1016/j.clnu.2022.10.024. Epub 2022 Nov 2. PMID 36502573
- [Background] Huang Q, Braffett BH, Simmens SJ, Young HA, Ogden CL. Dietary Polyphenol Intake in US Adults and 10-Year Trends: 2007-2016. J Acad Nutr Diet. 2020 Nov;120(11):1821-1833. doi: 10.1016/j.jand.2020.06.016. Epub 2020 Aug 15. PMID 32807722
- [Background] Kapolou, A. K. H. R., N; Koutelidakis, A. (2021). Association of Mean Daily Polyphenols Intake with Mediterranean Diet Adherence and Anthropometric Indices in Healthy Greek Adults: A Retrospective Study. Applied Sciences, 11(10). https://doi.org/10.3390/app11104664
- [Background] Ljotsson B, Jones M, Talley NJ, Kjellstrom L, Agreus L, Andreasson A. Discriminant and convergent validity of the GSRS-IBS symptom severity measure for irritable bowel syndrome: A population study. United European Gastroenterol J. 2020 Apr;8(3):284-292. doi: 10.1177/2050640619900577. Epub 2020 Jan 14. PMID 32213021
- [Background] Ma G., C., Y. (2020). Polyphenol supplementation benefits human health via gut microbiota: A systematic review via meta-analysis. . Journal of Functional Foods, 66(103829).
- [Background] Park SY, Kim YD, Kim MS, Kim KT, Kim JY. Cinnamon (Cinnamomum cassia) water extract improves diarrhea symptoms by changing the gut environment: a randomized controlled trial. Food Funct. 2023 Feb 6;14(3):1520-1529. doi: 10.1039/d2fo01835g. PMID 36655542
- [Background] Pietrzak A, Banasiuk M, Szczepanik M, Borys-Iwanicka A, Pytrus T, Walkowiak J, Banaszkiewicz A. Sodium Butyrate Effectiveness in Children and Adolescents with Newly Diagnosed Inflammatory Bowel Diseases-Randomized Placebo-Controlled Multicenter Trial. Nutrients. 2022 Aug 11;14(16):3283. doi: 10.3390/nu14163283. PMID 36014789
- [Background] Qaisar R, Iqbal MS, Ahmad F, Karim A. Oral butyrate improves postural balance by repairing leaky gut in geriatric adults. Gait Posture. 2025 Sep;121:370-376. doi: 10.1016/j.gaitpost.2025.06.016. Epub 2025 Jun 24. PMID 40577952
- [Background] Recharla N, Geesala R, Shi XZ. Gut Microbial Metabolite Butyrate and Its Therapeutic Role in Inflammatory Bowel Disease: A Literature Review. Nutrients. 2023 May 11;15(10):2275. doi: 10.3390/nu15102275. PMID 37242159
- [Background] Rosner, B. (2006). Hypothesis Testing Two-Sample INference. In Fundamentals of Biostatistics (6th ed., pp. 331-334). Duxbury Press.
- [Background] Wang X, Qi Y, Zheng H. Dietary Polyphenol, Gut Microbiota, and Health Benefits. Antioxidants (Basel). 2022 Jun 20;11(6):1212. doi: 10.3390/antiox11061212. PMID 35740109